CLINICAL TRIAL: NCT00829972
Title: Vitamin D Levels in Children Undergoing Adenotonsillectomies and Controls
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16687B
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: children undergoing adenotonsillectomy
- 2: children undergoing elective procedures other than adenotonsillectomy

SUMMARY:
The investigators aim to evaluate the levels of serum Vitamin D in children having their tonsils removed and appropriate controls. The investigators hypothesize that children undergoing tonsil removal will have lower Vit D levels than accepted norms and when compared to controls. The investigators also hypothesize that Vitamin D deficiency will correlate with indicators of inflammation such as C-Reactive Protein (CRP) and tonsil size.

ELIGIBILITY:
Inclusion Criteria:

* children age 1-12 undergoing adenotonsillectomy (active) or elective surgery such as hernia repair (control)

Exclusion Criteria:

* children on systemic steroids or multivitamins containing vitamin D
* control subjects with: a history of snoring, recurrent tonsillitis or score equal to or higher than 5 on the OSA questionnaire.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children age 1-12 years undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2009-09-01 (Actual); Study Completion 2009-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fuad M Baroody, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States